CLINICAL TRIAL: NCT07203118
Title: A Phase II/III Seamless Design Clinical Trial of Hepenofovir Fumarate Tablets (HTS) for Chronic Hepatitis B
Brief Title: A Phase II/III of Hepenofovir Fumarate Tablets (HTS) for Chronic Hepatitis B
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XAXT-2024-001
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HTS 20mg (Experimental)
  Interventions: Drug: HTS 20mg
- HTS 30mg (Experimental)
  Interventions: Drug: HTS 30mg
- HTS 40mg (Experimental)
  Interventions: Drug: HTS 40mg
- TAF 25mg (Experimental)
  Interventions: Drug: TAF 25mg

INTERVENTIONS:
Drug: HTS 20mg — Once daily, administered concomitantly with one TAF placebo tablet per dose, taken once daily with or within 30 minutes after a meal.
  Arms: HTS 20mg
Drug: HTS 30mg — Once daily, administered concomitantly with one TAF placebo tablet per dose, taken once daily with or within 30 minutes after a meal.
  Arms: HTS 30mg
Drug: HTS 40mg — Once daily, administered concomitantly with one TAF placebo tablet per dose, taken once daily with or within 30 minutes after a meal.
  Arms: HTS 40mg
Drug: TAF 25mg — Once daily, administered concomitantly with one HTS placebo tablet per dose, taken once daily with or within 30 minutes after a meal.
  Arms: TAF 25mg

SUMMARY:
UsingTAF as the control, the nvestigators aim to further explore the efficacy and safety of different dosages of HTS in the treatment of patients with chronic hepatitis B; ultimately, the nvestigators determine the optimal recommended dosage of HTS to provide a basis for Phase III confirmatory clinical research.

ELIGIBILITY:
Inclusion Criteria:

1）Age between 18 to 65 years old (inclusive), regardless of gender. 2) Meets diagnostic criteria for chronic hepatitis B (documented HBsAg positivity or HBV DNA positivity for more than 6 months, or confirmed by liver biopsy histopathology).

3)No prior treatment with any nucleos(t)ide analogue oral antiviral therapy; or, previous treatment with any nucleos(t)ide analogue must have ended at least 6 months prior to baseline.

4) Any interferon therapy (both pegylated and non-pegylated) must be completed at least 1 year prior to baseline visit.

5) Willing to use effective non-pharmacological contraception during the trial period.

Exclusion Criteria:

1. Hypersensitive to the study drug, its metabolites or any excipient in its formula;
2. With previous or present clinical hepatic decompensation (e.g., ascites, hepatic encephalopathy or varicose vein haemorrhage)
3. Complicated with liver diseases, including chronic alcoholic hepatitis, drug-induced hepatitis, etc.
4. Complicated with HCV, HIV or HDV infections
5. Documented resistance to the antiviral drug (Tenofovir).
6. Any cardiovascular, hematologic,pulmonary or nervous diseases deemed serious by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1444 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events of the Optimal Dosing Regimen as assessed by CTCAE v5.0 | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, changchun, China

IPD SHARING:
Plan to Share IPD: No